CLINICAL TRIAL: NCT01270503
Title: Meningococcal (Groups A, C, Y, W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®) Post-Marketing Safety Study in Healthy Children (2-11 Years), Adolescents (12-17 Years) and Adults (18-55 Years) in the Philippines
Brief Title: Post-Marketing Safety Study of Menactra® in Healthy Children, Adolescents, and Adults in the Philippines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA71; U1111-1116-4853 (Other: WHO)
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-10

CONDITIONS: Meningitis; Meningococcal Disease
Keywords: Meningitis; Meningococcal disease; Menactra®
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Menactra® Group 1 (Experimental): Participants aged 2 to 11 on enrollment
  Interventions: Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Menactra® Group 2 (Experimental): Participants aged 12 to 17 on enrollment
  Interventions: Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Menactra® Group 3 (Experimental): Participants aged 18 to 55 on enrollment
  Interventions: Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate

INTERVENTIONS:
Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Group 1
Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Group 2
Biological: Menactra®: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Group 3

SUMMARY:
This aim of the study is to assess post-marketing safety of a single dose of Menactra® vaccine with the intent to support conversion from monitored release to initial registration of Menactra® vaccine in the Philippines.

Primary Objective:

To describe the serious adverse events occurring within 30 days among participants who have received one dose of Menactra® vaccine.

DETAILED DESCRIPTION:
Each study participant will receive one dose of Menactra® vaccine and will be monitored for safety for 30 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 11 years of age on the day of inclusion (Group 1)
* Aged 12 to 17 years of age on the day of inclusion (Group 2)
* Aged 18 to 55 years of age on the day of inclusion (Group 3)
* Provision of informed consent form signed by the parent(s) or legal representative (Group 1)
* Provision of assent form signed by the subject and informed consent form signed by the parent (s) or legal representative (Group 2)
* Provision of informed consent form signed by the subject (Group 3)
* If the subject (Group 3) or the subject's parents or legally accepted representative (Group 1 and 2) are illiterate, an independent witness is required to sign the consent form
* Subject and parent/legally acceptable representative (if applicable) able to attend all scheduled visits and comply with all trial procedures
* For a woman of child-bearing potential, sexually active, use of a medically acceptable and effective method of contraception for at least 4 weeks prior to vaccination, until at least 4 weeks after vaccination (not applicable for females not of child-bearing potential or not sexually active).

Exclusion Criteria:

* For a woman of child-bearing potential sexually active, known or suspected pregnancy or positive serum/urine pregnancy test (not applicable for females not of child-bearing potential or not sexually active)
* Breast-feeding woman
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months or long-term systemic corticosteroid therapy
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or to a vaccine containing any of the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine during the present trial period
* Known personal or maternal Human Immunodeficiency virus (HIV), Hepatitis B antigen or Hepatitis C seropositivity as reported by the subject/parent/guardian and/or based on medical history
* History of seizures
* Thrombocytopenia, bleeding disorder or anticoagulants in the 3 weeks preceding inclusion contraindicating intramuscular injection
* Personal of family history of Guillain-Barré Syndrome.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 538 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Philippines, Inc.
Locations (127):
- Philippines (127):
  - General Santos, Antique
  - Calamba, Bataan
  - Marikina City, Batangas
  - Montalban, Batangas
  - Navotas, Batangas
  - Noveleta, Batangas
  - Olongapo City, Batangas
  - Paranaque City, Batangas
  - Pasay, Batangas
  - Pasig, Batangas
  - Plaridel, Batangas
  - Quezon City, Batangas
  - Angeles City, Benguet
  - Bacolod City, Benguet
  - Baguio City, Benguet
  - Baliwag, Benguet
  - Cagayan de Oro, Bulacan
  - Cardona, Bulacan
  - Cavite City, Bulacan
  - Cebu, Bulacan
  - Cebu, Capiz
  - City of Muntinlupa, Cavite
  - Naguila, Cavite
  - Olongapo City, Cavite
  - Ormoc City, Cavite
  - Ortigas, Cavite
  - Paranaque City, Cavite
  - Pasay, Cavite
  - Pasig, Cavite
  - Pulilan, Cavite
  - Quezon City, Cavite
  - Quezon City, Cebu
  - Roxas, Cebu
  - San Fernando City, Cebu
  - San Jose, Cebu
  - Santa Rosa, Cebu
  - Tagug, Davao Del Norte
  - City of Taguig, Davao Del Sur
  - Santa Rosa, Davao Del Sur
  - Tacloban City, Davao Del Sur
  - Talisay City, Davao Del Sur
  - Tarlac City, Davao Del Sur
  - Taytay, Davao Del Sur
  - Theresa, Davao Del Sur
  - Valenzuela, Davao Del Sur
  - Bacolod City, Ilocos Norte
  - Baguio City, Ilocos Norte
  - Dasmariñas, Iloilo
  - General Santos, Iloilo
  - Iloilo City, Iloilo
  - Angeles City, Isabela
  - Baguio City, Isabela
  - Alaminos, LA Union
  - Bacolod City, La Union
  - City of Muntinlupa, Laguna
  - Ormoc City, Laguna
  - Quezon City, Laguna
  - Tacloban City, Lanao Del Norte
  - Tanauan, Lanao Del Norte
  - Quezon City, Leyte
  - San Fernando City, Leyte
  - San Miguel, Leyte
  - City of Taguig, Misamis Oriental
  - Santa Rosa, Misamis Oriental
  - Tarlac City, Misamis Oriental
  - Batangas, NCR
  - Bocaue, NCR
  - Cabanatuan City, NCR
  - Calamba, NCR
  - Caloocan, NCR
  - Cebu, NCR
  - Concepcion, NCR
  - Dagupan, NCR
  - Dasmariñas, NCR
  - Davao City, NCR
  - Fairview, NCR
  - Guagua, NCR
  - Iligan City, NCR
  - Iloilo City, NCR
  - Imus, NCR
  - Kidapawan, NCR
  - La Trinidad, NCR
  - Laoag, NCR
  - Las Piñas, NCR
  - Lipa, NCR
  - Lipa City, NCR
  - Los Baños, NCR
  - Maasin, NCR
  - Makati, NCR
  - Makati City, NCR
  - Malabon, NCR
  - Malolos, NCR
  - Mandaluyong, NCR
  - Quezon City, Negros Occidental
  - Roxas City, Negros Occidental
  - San Fernando City, Negros Occidental
  - San Jose del Monte, Negros Occidental
  - Urdaneta, North Cotobato
  - Manila, NRC
  - Marikina City, NRC
  - Baguio City, Nueva Ecija
  - Batangas, Pampanga
  - Biñan, Pampanga
  - Cagayan de Oro, Pampanga
  - Caloocan, Pampanga
  - Cebu, Pampanga
  - Angeles City, Pangasinan
  - Bacoor, Pangasinan
  - Baguio City, Pangasinan
  - Balanga, Pangasinan
  - Imus, Pasig City
  - Concepcion, Rizal
  - Davao City, Rizal
  - General Santos, Rizal
  - Imus, Rizal
  - Tacloban City, South Cotabato
  - Tagum, South Cotabato
  - Tanauan, South Cotabato
  - Tarlac City, South Cotabato
  - Taytay, South Cotabato
  - San Pedro, Southern Leyte
  - Angeles City, Tarlac
  - Bacolod City, Tarlac
  - Baguio City, Tarlac
  - Batangas, Zambales
  - Calamba, Zambales
  - Cauayan, Zambales

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 16 December 2010 through 15 November 2012 at 130 clinic centers in thePhillipines
Pre-assignment Details: A total of 538 participants who met all of the inclusion and none of the exclusion criteria were vaccinated in this study.
Groups:
- Menactra® Vaccine Group: Participants who received a single dose of Menactra vaccine
Period: Overall Study
Arm/Group | Menactra® Vaccine Group
Started | 538
Completed | 537
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 538
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 468
  Between 18 and 65 years | 70
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 9.3 (10.3)
Gender [Number; unit: participants] — Gender information was missing for 3 participants in the study
  participants
    Female | 272
    Male | 263
Region of Enrollment [Number; unit: Participants]
  Philippines | 538

OUTCOME MEASURES:

1. Primary Outcome: Safety Overview Within 30 Days in Participants Vaccinated With Menactra®
Time Frame: Day 0 up to Day 30 post-vaccination
Population: Post-vaccination safety were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 537
Participants
  Serious adverse event | 0
  Non-serious related adverse event not listed in PI | 2

2. Secondary Outcome: Number of Subjects Reporting Non-serious Related Adverse Events Not Listed in Prescribing Information (PI) Following Vaccination With Menactra®
Time Frame: Day 0 up to Day 30 post-vaccination
Population: Post-vaccination safety were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Groups:
- Menactra® Vaccine Group: Participants received a single dose of Menactra vaccine
Arm/Group | Menactra® Vaccine Group
Number analyzed (Participants) | 537
Participants
  Pyrexia | 2
  Other non-serious related adverse events | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post vaccination) up to Day 30 post vaccination.
Arm/Group | Menactra® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/538
Other Adverse Events (participants affected / at risk) | 0/537

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications